CLINICAL TRIAL: NCT00169624
Title: The DIAMET Study: Peripheral and Coronary Endothelial Dysfunction in Type 2diabetic Patients- Evaluation of Reversibility Following 3 Months of Metformin Treatment
Brief Title: Peripheral and Coronary Endothelial Dysfunction In Type 2diabetic Patients- Role of Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2004.346
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Coronary and Peripheral Endothelial Dysfunction
Keywords: Diabetes,; coronary endothelial dysfunction,; metformin,; glyclazide,; MRI.
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; Gliclazide

INTERVENTIONS:
Drug: Metformin
Drug: Gliclazide

SUMMARY:
Peripheral and coronary endothelial dysfunction in type 2 diabetic patients may be influenced by therapeutics. Using Radial flow monitoring and myocardial perfusion magnetic resonance imaging, we designed a controlled randomized double blind study to test the hypothesis that endothelial dysfunction will be reversed following 3 months of Metformin administration vs gliclazide. 30 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

18-70 years old, type 2 diabetes, non significant coronary atherosclerosis on inclusion coronary angiogram (ie no coronary stenosis > 70%), HbA1c<9%

Exclusion Criteria:

significant coronary stenosis (>70%), lack of informed consent, unstable hypertension, renal failure, contra-indication to metformin or gliclazide, pregnancy, atrial fibrillation, contraindication to MRI, or to adenosine, brachial artery calcifications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10

PRIMARY OUTCOMES:
Flow dependent and independent Brachial artery vasoreactivity assessed using Doppler technology at 3 month vs baseline

SECONDARY OUTCOMES:
Myocardial perfusion improvement following improved vasoreactivity assessed using myocardial perfusion imaging at 3 month vs baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SEBBAG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Laurent SEBBAG, Lyon, France